CLINICAL TRIAL: NCT05891535
Title: Stentless Florence Robotic Intracorporeal Neobladder (FloRIN)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Luca Lambertini, Professor, University of Florence
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StentlessFloRIN
Record Dates: First submitted 2023-05-24; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Perioperative Complication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stentless FloRIN (Experimental): Florence robotic Intra Corporeal Neobladder configuration was performed without the employement of Mono J ureteral catheters
  Interventions: Procedure: Robot assisted radical cystectomy without mono J ureteral stent placement
- Stented FloRIN (Active Comparator): Florence robotic Intra Corporeal Neobladder configuration was performed with the employement of Mono J ureteral catheters
  Interventions: Procedure: Robot assisted radical cystectomy with mono J ureteral stent placement

INTERVENTIONS:
Procedure: Robot assisted radical cystectomy without mono J ureteral stent placement — Robot assisted radical cystectomy with/without ureteral mono J stent placement during uretero-neobladder anastomosis
  Arms: Stentless FloRIN
Procedure: Robot assisted radical cystectomy with mono J ureteral stent placement — Robot assisted radical cystectomy with/without ureteral mono J stent placement during uretero-neobladder anastomosis
  Arms: Stented FloRIN

SUMMARY:
Objective: To investigate perioperative and mid-term functional outcomes of stentless FloRIN reconfiguration as compared to standard technique performed with ureteral mono J placement.

Patient and dataset Clinical and surgical data of all consecutive patients treated at our Institution from January 2021 to February 2022 with RARC, lymph node dissection (LND) and FloRIN reconfiguration were gathered in this single institution randomized 1:1 prospective series. All patients with clinical stage T1-T4N0-N1M0 amenable to radical cystectomy with curative intent and FloRIN reconfiguration were included. The sample size for a non-inferiority trial was calculated for different endpoints. Preoperative work-up included chest and abdomen contrast-enhanced computed tomography (CT) scan. Main exclusion criteria were: 1) presence of one or multiple tumor metastases at preoperative staging; 2) histopathological confirmation of bladder tumor at the level of prostatic urethra; 3) treatment without curative intent (cT4b, salvage or palliative cystectomies); 4) presence of urethral stricture. After preliminary multidisciplinary evaluation, patients were randomly assigned with 1:1 ratio to the mono-J stent placement or the stentless group. For the present study, only patients with a minimum 6 month-follow up were evaluated. Patient demographics, including ASA score and Charlson Comorbidity Index (CCI), peri- and postoperative features including operative time, conversion rate, estimated blood loss (EBL), Visual Analogue Scale (VAS) pain intensity scale, length of hospital stay (LOS) early (≤30 days) and delayed (>30 days) complications rate, and pathological data were thoroughly gathered.

Follow-up schedule included blood analysis and CT scan performed three months after surgery, then every 6 months from the first to the third postoperative year, followed by annual imaging assessment according to individual risk profile, as postulated by the EAU guidelines. In case of newly diagnosed postoperative hydronephrosis, only patients with grade > 2 or symptomatic were assessed as functional failure. All eligible patients were offered the possibility to undergo neoadjuvant cisplatin-based chemotherapy before RARC. Patients with non-muscle invasive bladder cancer, cN+ disease and those presenting with severe cardiovascular morbidity or high preoperative creatinine levels, strongly contraindicating cisplatin administration, underwent immediate radical cystectomy. The enhanced recovery after surgery protocol (ERAS) was regularly applied. Suitable patients underwent a nutritional assessment with a specific immune-nutrition, 7 days preoperatively.

DETAILED DESCRIPTION:
Surgical technique All robotic surgical procedures were performed by a single highly experienced robotic surgeon (AM) alternated with the other fellow-members. The Da Vinci Si system, (Intuitive Surgical, Sunnyvale, CA, USA), in a four-arm conﬁguration with a 0/30° laparoscope was used for all cases. As previously described (4), patients are positioned in 30° Trendelenburg with a standard six-port transperitoneal approach for the demolitive part and then reduced to 20° to facilitate bowel handling and urethro-neobladder anastomosis. After the isolation of 45-50 cm of ileum, the urethro-ileal anastomosis is performed obtaining an asymmetrical 'U'-shape (25-30 cm distally and 20 cm proximally to anastomosis). Ileum is then sectioned by endo- GIA 60 mm Echelon Powered Endopath Stapler (Ethicon Inc., Cincinnati, OH, USA) and the intestinal continuity is then restored with an intracorporeal side-to-side anastomosis with one longitudinal fire. The two transversal holes are closed by a double layer 3-0 Stratafix running suture. The asymmetrical 'U'-shape segment is then detubularized and the posterior plate is reconfigured as an "Γ", by suturing the span of the arms of the 'U' aligned in parallel, and by placing the extending portion of the loop distally to the right, forming the short arm of the "Γ". Neobladder neck configuration was performed by suturing a tract of 2-5 cm longitudinally from the 12 o'clock position of the anastomosis. Then, the posterior plate was folded anteriorly, distal to proximally, roughly 5 cm right from the proximal edge of the posterior closure with the goal of creating two symmetrical segments.

Ureteral reimplantation After a careful isolation of the ureters avoiding iatrogenic blood supply damages, the ureteric stumps were sectioned and adequately spatulated. Bilateral ureteral reimplantation was then performed orthotopically and directly with no anti-reflux mechanisms on the lateral side of each anterior segment with mucosa-mucosa inverted sutures. In case of stentless procedure the anastomosis was performed directly while mono J ureteral catheters were employed in case of stent placement. The anterior plate was therefore closed by an "∧" -shaped suture. Both mono J stents were passed through the closing of the two anterior plates in the stent group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed Bladder Cancer with clinical stage T1-T4N0-N1M0
* Patients amenable to radical cystectomy with eligible to orthotopic neobladder reconfiguration curative intent and FloRIN reconfiguration were included.

Exclusion Criteria:

* Presence of one or multiple tumor metastases at preoperative staging
* Histopathological confirmation of bladder tumor at the level of prostatic urethra; - Treatment without curative intent (cT4b, salvage or palliative cystectomies)
* Presence of urethral stricture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Mid term complications | 6 months
  Mid term complications rate

SECONDARY OUTCOMES:
Preoperative complications | 7 days
  Perioperative complications rate

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Minervini, Prof., Study Director — University of Florence
Locations (1):
- Careggi hospital, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed K, Khan SA, Hayn MH, Agarwal PK, Badani KK, Balbay MD, Castle EP, Dasgupta P, Ghavamian R, Guru KA, Hemal AK, Hollenbeck BK, Kibel AS, Menon M, Mottrie A, Nepple K, Pattaras JG, Peabody JO, Poulakis V, Pruthi RS, Redorta JP, Rha KH, Richstone L, Saar M, Scherr DS, Siemer S, Stoeckle M, Wallen EM, Weizer AZ, Wiklund P, Wilson T, Woods M, Khan MS. Analysis of intracorporeal compared with extracorporeal urinary diversion after robot-assisted radical cystectomy: results from the International Robotic Cystectomy Consortium. Eur Urol. 2014 Feb;65(2):340-7. doi: 10.1016/j.eururo.2013.09.042. Epub 2013 Oct 9. PMID 24183419
- [Background] Dell'Oglio P, Mazzone E, Lambert E, Vollemaere J, Goossens M, Larcher A, Van Der Jeugt J, Devos G, Poelaert F, Uvin P, Collins J, De Naeyer G, Schatteman P, D'Hondt F, Mottrie A. The Effect of Surgical Experience on Perioperative and Oncological Outcomes After Robot-assisted Radical Cystectomy with Intracorporeal Urinary Diversion: Evidence from a Referral Centre with Extensive Experience in Robotic Surgery. Eur Urol Focus. 2021 Mar;7(2):352-358. doi: 10.1016/j.euf.2020.01.016. Epub 2020 Feb 13. PMID 32061537
- [Background] McCulloch P, Altman DG, Campbell WB, Flum DR, Glasziou P, Marshall JC, Nicholl J; Balliol Collaboration; Aronson JK, Barkun JS, Blazeby JM, Boutron IC, Campbell WB, Clavien PA, Cook JA, Ergina PL, Feldman LS, Flum DR, Maddern GJ, Nicholl J, Reeves BC, Seiler CM, Strasberg SM, Meakins JL, Ashby D, Black N, Bunker J, Burton M, Campbell M, Chalkidou K, Chalmers I, de Leval M, Deeks J, Ergina PL, Grant A, Gray M, Greenhalgh R, Jenicek M, Kehoe S, Lilford R, Littlejohns P, Loke Y, Madhock R, McPherson K, Meakins J, Rothwell P, Summerskill B, Taggart D, Tekkis P, Thompson M, Treasure T, Trohler U, Vandenbroucke J. No surgical innovation without evaluation: the IDEAL recommendations. Lancet. 2009 Sep 26;374(9695):1105-12. doi: 10.1016/S0140-6736(09)61116-8. PMID 19782876
- [Background] Minervini A, Vanacore D, Vittori G, Milanesi M, Tuccio A, Siena G, Campi R, Mari A, Gavazzi A, Carini M. Florence robotic intracorporeal neobladder (FloRIN): a new reconfiguration strategy developed following the IDEAL guidelines. BJU Int. 2018 Feb;121(2):313-317. doi: 10.1111/bju.14077. Epub 2017 Dec 11. PMID 29140596
- [Background] Di Maida F, Grosso AA, Tasso G, Gemma L, Lambertini L, Nardoni S, Mari A, Tuccio A, Vittori G, Masieri L, Minervini A. Robot assisted radical cystectomy with Florence Robotic Intracorporeal Neobladder (FloRIN): Functional and urodynamic features compared with a contemporary series of open Vescica Ileale Padovana (VIP). Eur J Surg Oncol. 2022 Aug;48(8):1854-1861. doi: 10.1016/j.ejso.2022.04.007. Epub 2022 Apr 20. PMID 35484043
- [Background] Minervini A, Di Maida F, Tasso G, Mari A, Bossa R, Sforza S, Grosso AA, Tellini R, Vittori G, Siena G, Tuccio A, Masieri L, Carini M. Robot assisted radical cystectomy with Florence robotic intracorporeal neobladder (FloRIN): Analysis of survival and functional outcomes after first 100 consecutive patients upon accomplishment of phase 3 IDEAL framework. Eur J Surg Oncol. 2021 Oct;47(10):2651-2657. doi: 10.1016/j.ejso.2021.05.007. Epub 2021 May 15. PMID 34023169
- [Background] Beano H, He J, Hensel C, Worrilow W, Townsend W, Gaston K, Clark PE, Riggs S. Safety of decreasing ureteral stent duration following radical cystectomy. World J Urol. 2021 Feb;39(2):473-479. doi: 10.1007/s00345-020-03191-2. Epub 2020 Apr 17. PMID 32303901
- [Background] Scotland KB, Lo J, Grgic T, Lange D. Ureteral stent-associated infection and sepsis: pathogenesis and prevention: a review. Biofouling. 2019 Jan;35(1):117-127. doi: 10.1080/08927014.2018.1562549. Epub 2019 Feb 8. PMID 30732463
- [Background] Peng YL, Ning K, Wu ZS, Li ZY, Deng MH, Xiong LB, Yu CP, Zhang ZL, Liu ZW, Lu HM, Zhou FJ. Ureteral stents cannot decrease the incidence of ureteroileal anastomotic stricture and leakage: A systematic review and meta-analysis. Int J Surg. 2021 Sep;93:106058. doi: 10.1016/j.ijsu.2021.106058. Epub 2021 Aug 18. PMID 34416355
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Joyce CR, Zutshi DW, Hrubes V, Mason RM. Comparison of fixed interval and visual analogue scales for rating chronic pain. Eur J Clin Pharmacol. 1975 Aug 14;8(6):415-20. doi: 10.1007/BF00562315. PMID 1233242
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Witjes JA, Bruins HM, Cathomas R, Comperat EM, Cowan NC, Gakis G, Hernandez V, Linares Espinos E, Lorch A, Neuzillet Y, Rouanne M, Thalmann GN, Veskimae E, Ribal MJ, van der Heijden AG. European Association of Urology Guidelines on Muscle-invasive and Metastatic Bladder Cancer: Summary of the 2020 Guidelines. Eur Urol. 2021 Jan;79(1):82-104. doi: 10.1016/j.eururo.2020.03.055. Epub 2020 Apr 29. PMID 32360052
- [Background] Stangl-Kremser J, Lambertini L, Di Maida F, Martinez-Fundichely A, Ferro M, Pradere B, Soria F, Albisinni S, Wu Z, Del Giudice F, Cacciamani GE, Valerio M, Briganti A, Roupret M, Shariat SF, Lee C, Minervini A, Moschini M, Mari A; European Association of Urology-Young Academic Urologists Urothelial Carcinoma Working Group. Enhancing Recovery After Major Bladder Cancer Surgery: Comprehensive Review and Assessment of Application of the Enhanced Recovery After Surgery Guidelines. Eur Urol Focus. 2022 Nov;8(6):1622-1626. doi: 10.1016/j.euf.2022.06.004. Epub 2022 Jun 27. PMID 35773181
- [Background] Hussein AA, Elsayed AS, Aldhaam NA, Jing Z, Peabody JO, Wijburg CJ, Wagner A, Canda AE, Khan MS, Scherr D, Schanne F, Maatman TJ, Kim E, Mottrie A, Aboumohamed A, Gaboardi F, Pini G, Kaouk J, Yuh B, Rha KH, Hemal A, Palou Redorta J, Badani K, Saar M, Stockle M, Richstone L, Roupret M, Balbay D, Dasgupta P, Menon M, Guru KA. A comparative propensity score-matched analysis of perioperative outcomes of intracorporeal vs extracorporeal urinary diversion after robot-assisted radical cystectomy: results from the International Robotic Cystectomy Consortium. BJU Int. 2020 Aug;126(2):265-272. doi: 10.1111/bju.15083. Epub 2020 May 16. PMID 32306494
- [Background] Mastroianni R, Ferriero M, Tuderti G, Anceschi U, Bove AM, Brassetti A, Misuraca L, Zampa A, Torregiani G, Ghiani E, Giannarelli D, Guaglianone S, Gallucci M, Simone G. Open Radical Cystectomy versus Robot-Assisted Radical Cystectomy with Intracorporeal Urinary Diversion: Early Outcomes of a Single-Center Randomized Controlled Trial. J Urol. 2022 May;207(5):982-992. doi: 10.1097/JU.0000000000002422. Epub 2022 Feb 2. PMID 34986007
- [Background] Cacciamani GE, De Marco V, Sebben M, Rizzetto R, Cerruto MA, Porcaro AB, Gill IS, Artibani W. Robot-assisted Vescica Ileale Padovana: A New Technique for Intracorporeal Bladder Replacement Reproducing Open Surgical Principles. Eur Urol. 2019 Sep;76(3):381-390. doi: 10.1016/j.eururo.2018.11.037. Epub 2018 Nov 30. PMID 30509764
- [Background] Balbay MD, Canda AE, Kiremit MC, Koseoglu E. Intracorporeal Studer Pouch Formation with Balbay's Technique Following Robotic Radical Cystectomy for Bladder Cancer: Experience with 22 Cases with Oncologic and Functional Outcomes. J Endourol. 2020 Mar;34(3):273-280. doi: 10.1089/end.2019.0559. Epub 2020 Mar 3. PMID 31731881
- [Background] Tan WP, Whelan P, Deane LA. Intentional Omission of Ureteral Stents During Robotic-assisted Intracorporeal Ureteroenteric Anastomosis: Is It Safe and Feasible? Urology. 2017 Apr;102:116-120. doi: 10.1016/j.urology.2017.01.014. Epub 2017 Jan 19. PMID 28111222
- [Background] Ramahi YO, Shiekh M, Shah AA, Houenstein H, Ely HB, Shabir U, Jing Z, Li Q, Hussein AA, Guru KA. Uretero-enteric Strictures After Robot Assisted Radical Cystectomy: Prevalence and Management Over Two Decades. Clin Genitourin Cancer. 2023 Apr;21(2):e19-e26. doi: 10.1016/j.clgc.2022.10.006. Epub 2022 Oct 12. PMID 36372690
- [Background] Carbonara U, Crocerossa F, Mehrazin R, Campi R, Marchioni M, Morlacco A, Paglairulo V, Wu Z, Autorino R, Stein RJ, Eun D, Ditonno P, Dal Moro F. Robotic ureteral reimplantation: systematic review and pooled analysis of comparative outcomes in adults. Minerva Urol Nephrol. 2022 Apr;74(2):161-168. doi: 10.23736/S2724-6051.21.04558-4. Epub 2022 Feb 11. PMID 35147383
- [Background] Wilson TG, Guru K, Rosen RC, Wiklund P, Annerstedt M, Bochner BH, Chan KG, Montorsi F, Mottrie A, Murphy D, Novara G, Peabody JO, Palou Redorta J, Skinner EC, Thalmann G, Stenzl A, Yuh B, Catto J; Pasadena Consensus Panel. Best practices in robot-assisted radical cystectomy and urinary reconstruction: recommendations of the Pasadena Consensus Panel. Eur Urol. 2015 Mar;67(3):363-75. doi: 10.1016/j.eururo.2014.12.009. Epub 2015 Jan 9. PMID 25582930
- [Background] Tomer N, Garden E, Small A, Palese M. Ureteral Stent Encrustation: Epidemiology, Pathophysiology, Management and Current Technology. J Urol. 2021 Jan;205(1):68-77. doi: 10.1097/JU.0000000000001343. Epub 2020 Aug 28. PMID 32856981
- [Background] Aldhaam NA, Hussein AA, Elsayed AS, Jing Z, Osei J, Kurbiel Z, Babar T, Khan S, Nagra A, Segal B, Li Q, Guru KA. Detailed Analysis of Urinary Tract Infections After Robot-Assisted Radical Cystectomy. J Endourol. 2021 Jan;35(1):62-70. doi: 10.1089/end.2020.0316. Epub 2020 Nov 6. PMID 32664741
- [Background] Sasaki Y, Takahashi M, Fukuta K, Shiozaki K, Daizumoto K, Ozaki K, Ueno Y, Tsuda M, Kusuhara Y, Fukawa T, Yamamoto Y, Yamaguchi K, Izaki H, Kanda K, Kanayama H. The patient-side surgeon plays a key role in facilitating robot-assisted intracorporeal ileal conduit urinary diversion in men. J Robot Surg. 2022 Apr;16(2):437-444. doi: 10.1007/s11701-021-01256-x. Epub 2021 Jun 3. PMID 34081290
- [Background] Tan TW, Nair R, Saad S, Thurairaja R, Khan MS. Safe transition from extracorporeal to intracorporeal urinary diversion following robot-assisted cystectomy: a recipe for reducing operative time, blood loss and complication rates. World J Urol. 2019 Feb;37(2):367-372. doi: 10.1007/s00345-018-2386-4. Epub 2018 Jun 22. PMID 29934671